CLINICAL TRIAL: NCT00814138
Title: Phase II Trial of Methotrexate in Myasthenia Gravis
Brief Title: Efficacy of Methotrexate in Myasthenia Gravis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Richard Barohn, MD, Gertrude and Dewey Zeigler Professor of Neurology, Chairman Deptartment of Neurology, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11552; FDA OOPD 003538 (Other Grant/Funding Number: RO1FD003538)
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Myasthenia Gravis
Keywords: myasthenia gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Methotrexate
  Interventions: Drug: Methotrexate
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Methotrexate — 10 mg weekly for 2 weeks and then increase to 15mg for 2 weeks and then 20mg weekly until the end of the study
  Arms: 1
Other: Placebo — Weekly
  Arms: 2

SUMMARY:
Myasthenia gravis is a rare neuromuscular disorder characterized by weakness and fatigability of ocular, bulbar, and extremity musculature. The specific aim of this study is to determine if oral methotrexate is an effective therapy for myasthenia gravis (MG) patients who are prednisone dependent. Patients will be randomized to receive either methotrexate or placebo and those who are entered onto this trial will have symptoms and signs of the disease while on prednisone therapy. The hypothesis is that adding methotrexate therapy in these patients will improve the MG manifestations so that the prednisone dose can be reduced and clinical measures of MG severity will improve.

Funding Source - FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

* Patients must have MGFA MG grades 2, 3, or 4 generalized myasthenia gravis, according to the MGFA classification system
* Elevated acetylcholine receptor antibody (AChR-Ab) titer.
* Patient's signs and symptoms should not be better explained by another disease process.
* Prednisone dose of at least 10 mg/day (or the equivalent in alternate days) and the subject must be on a stable dose of prednisone for 30 days prior to the screening visit.

Exclusion Criteria:

* A history of chronic degenerative, psychiatric, or neurologic disorder other than MG that can produce weakness or fatigue.
* Other major chronic or debilitating illnesses within six months prior to study entry.
* Female patients who are premenopausal and are: (a) pregnant on the basis of a serum pregnancy test, (b) breast-feeding, or (c) not using an effective method of double barrier (1 hormonal plus 1 barrier method or 2 simultaneous barrier methods) birth control (birth control pills, male condom, female condom, intrauterine device, Norplant, tubal ligation, or other sterilization procedures).
* Altered levels of consciousness, dementia, or abnormal mental status.
* Evidence of thymoma on chest CT or MRI. Such a finding could require immediate thymectomy and would preclude entry into the study.
* Thymectomy in the previous three months.
* Patients who have been medicated with azathioprine, cyclosporine, cyclophosphamide, mycophenolate mofetil, IVIg, or other immunosuppressive drugs within the last 60 days.
* Chest X-ray with evidence of tumor, infection, or interstitial lung disease.
* Clinical history of chronic or recurrent infections.
* Daily use of non-steroidal anti-inflammatory drugs (NSAIDs).
* History of renal or hepatic insufficiency or liver enzymes greater than the upper limit of normal.
* History of bone marrow hypoplasia, leucopenia, thrombocytopenia, significant anemia, clinical or laboratory evidence of immunodeficiency syndromes.
* Forced Vital Capacity (FVC) <50% of predicted.
* MG Grade 1 (ocular only) or 5 (crisis, requiring ventilator).
* Prior use of methotrexate for any condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Barohn, MD, Principal Investigator — University of Kansas Medical Center
Locations (16):
- United States (15):
  - Phoenix Neurological Associates, Phoenix, Arizona
  - University of California, San Francisco, Fresno, California
  - University of California-Irvine, Irvine, California
  - Forbes Norris MDA/ALS Research Center, San Francisco, California
  - University of Florida, Health Science Center Jacksonville, Jacksonville, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospitals, Boston, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Penn State College of Medicine, The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The Nerve and Muscle Center of Texas, Houston, Texas
  - University Health Sciences Center, San Antonio, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
- University of Toronto, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 - Methotrexate (2.5 mg): Methotrexate: 10 mg weekly for 2 weeks and then increase to 15mg for 2 weeks and then 20mg weekly until the end of the study
- Placebo: Placebo: 10 mg weekly for 2 weeks and then increase to 15mg for 2 weeks and then 20mg weekly until the end of the study
Period: Overall Study
Arm/Group | 1 - Methotrexate (2.5 mg) | Placebo
Started | 25 | 25
Completed | 24 | 18
Not Completed | 1 | 7

BASELINE CHARACTERISTICS:
Population: Eligible participatns were aged at least 18 years; had a diagnosis of generalized Myasthenia Gravis Foundation of America class II, III or IV; positive acetylcholine receptor antibodies; stable dose of greater than or equal to 10 mg/day of prednisone.
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 23
  >=65 years | 12 | 15 | 27
Age, Continuous [Mean (Full Range); unit: years] | 66.5 [28.5 to 83.9] | 68.6 [26.6 to 87.2] | 67.6 [26.6 to 87.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 19 | 16 | 35
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 4 | 7
  United States | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Total Prednisone Dose Area Under the Curve
Description: The primary outcome measure was the nine-month prednisone area under the dose-time curve (AUDTC, months 4-12). The AUDTC was chosen because it accounted for changes in the prednisone dose that could occur frequently during a month.
Time Frame: 9 months
Population: Myasthenia Gravis patients aged 18 and older that were acetylcholine antibody positive with a myasthenia gravis foundation score of Grade II, III or IV.
Measure: Number (95% Confidence Interval); unit: mg*Months
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 25 | 25
mg*Months | 2996.6 [1495.9 to 4497.3] | 3484.7 [2151.8 to 4817.5]
Statistical Analysis 1: Comparison: Methotrexate vs Placebo; If a study participant terminated, their last results were pulled forward; Test type: Superiority or Other; p = 0.26, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -488.0, 95% CI 2-sided [-2443.4 to 1467.3]

2. Secondary Outcome: Average Prednisone Daily Dose (mg/Day)
Description: Participants were asked to fill out the amount of prednisone they took every day on a paper diary.
Time Frame: Total length of time daily dose information was collected, i.e. 9 months.
Measure: Mean (95% Confidence Interval); unit: mg/day
Groups:
- Methotrexate: Methotrexate: 10 mg/day for 2 weeks and then increase to 15mg/day for 2 weeks and then 20mg/day until the end of the study
- Placebo: Placebo: 10 mg/day for 2 weeks and then increase to 15mg/day for 2 weeks and then 20mg/day until the end of the study
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 25 | 25
mg/day | 12.8 [9.1 to 16.5] | 14.6 [11.5 to 17.8]
Statistical Analysis 1: Comparison: Methotrexate vs Placebo; If a study participant terminated, their last results were pulled forward; Test type: Superiority or Other; p = 0.26, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-9.7 to 5.8]

3. Secondary Outcome: Quantitative Myasthenia Gravis (QMG) Score
Description: The QMG is a 13 item ordinal scale which measures ocular, bulbar, extremity fatigue and strength, along with respiratory function. The scale is from 0 - 3 for each item, with 0 meaning normal and 3 is severe. Total score can range from 0 to 39.
Time Frame: Change from Baseline to Month 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale | -1.4 [-2.9 to 0.1] | 0.3 [-1.8 to 2.4]
Statistical Analysis 1: Comparison: Methotrexate vs Placebo; If a study participant terminated, their last results were pulled forward; Test type: Superiority or Other; p = 0.29, t-test, 2 sided; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-4.9 to 1.5]

4. Secondary Outcome: Manual Muscle Testing 12 Month Change
Description: This measurement was developed to measure the strength of muscle groups in the face, neck, arms and legs. Measurement is made by grading the amount of weakness. Participants are graded as having normal, mild (25%) weakness, moderate (50%) weakness or severe (75%) weakness and 4 = paralyzed/unable to do. Normal would receive a score of 0, mild would receive a score of 1, moderate would receive a score of 2, severe would receive a score of 3 and unable to perform would receive a score of 4. Range would be from 0 (no weakness) to 76 (complete paralysis).
Time Frame: Change from Baseline to Month 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale | -5.5 [-7.4 to -3.8] | -3.3 [-6.6 to 0.1]
Statistical Analysis 1: Comparison: Methotrexate vs Placebo; If a study participant terminated, their last results were pulled forward; Test type: Superiority or Other; p = 0.28, t-test, 2 sided; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-6.3 to 1.8]

5. Secondary Outcome: MGQOL 12 Month Change
Description: This test is a 15 item patient-reported scale indicating how myasthenia gravis affects the quality of life. Each item is graded as how true each statement has been over the past 7 days. The scale is 0=Not at all, 1= a little bit, 2= somewhat, 3= quite a bit and 4= very much. The numbers are then added to produce a total score. The MGQOL score would range from 0 (no MG symptoms that affected their quality of life) to a score of 60 (MG symptoms affected they quality of life very much).
Time Frame: Change from Baseline to Month 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale | -4.6 [-9.1 to -0.1] | -3.7 [-8.4 to 1.0]
Statistical Analysis 1: Comparison: Methotrexate vs Placebo; If a study participant terminated, their last results were pulled forward; Test type: Superiority or Other; p = 0.82, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-7.2 to 5.4]

6. Secondary Outcome: MG-ADL 12 Month Change
Description: The MG-ADL is an 8 item scale developed to assess myasthenia gravis symptoms. Score will range from 0 (normal - no MG symptoms) to 24 (severe MG symptoms)
Time Frame: Change from Baseline to Month 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale | -1.2 [-2.3 to -0.5] | 0.26 [-0.9 to 1.5]
Statistical Analysis 1: Comparison: Methotrexate vs Placebo; If a study participant terminated, their last results were pulled forward; Test type: Superiority or Other; p = 0.21, t-test, 2 sided; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-3.7 to 0.8]

7. Secondary Outcome: MG Composite Change Over 12 Months
Description: This scale is composed of components of the QMG, MG-ADL and the MMT. These components have been shown to be the most responsive in previous clinical trials. Each item in the QMG, MG-ADL and the MMT was weighed (Rasch analysis performed) and then assigned a score. Score would range from 0 (no effects from the myasthenia gravis) to a score of 50. A participant with a score of 50 wwould be in the hospital on a ventilator.
Time Frame: Change from Baseline to Month 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale | -4.6 [-6.4 to -2.7] | -1.3 [-3.7 to 1.1]
Statistical Analysis 1: Comparison: Methotrexate vs Placebo; If a study participant terminated, their last results were pulled forward; Test type: Superiority or Other; p = 0.09, t-test, 2 sided; Mean Difference (Final Values) = -3.3, 95% CI 2-sided [-7.1 to 0.5]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the 12 months the participants participated in the study.
Groups:
- Methotrexate Group - Adverse Events: Reported the number of adverse events in the group randomized to methotrexate.
- Placebo Group - Adverse Events: Reported the number of adverse events in the group randomized to placebo
Arm/Group | Methotrexate Group - Adverse Events | Placebo Group - Adverse Events
Serious Adverse Events (participants affected / at risk) | 2/25 | 1/25
Other Adverse Events (participants affected / at risk) | 23/25 | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methotrexate Group - Adverse Events (N=25) | Placebo Group - Adverse Events (N=25)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) — Subject died after suffering a stroke at month 10. This was reviewed by the safety monitor and deemed not study medication related.
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject admitted to hospital for Pancreatitis. Determined to not be study medication related.
Thrombosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Subject was admitted to the hospital for possible thrombosis.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Participant admitted to the hospital for shortness of breath. This occurred between the screening visit and the baseline visit; therefore no medication had been dispensed at that time.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methotrexate Group - Adverse Events (N=25) | Placebo Group - Adverse Events (N=25)
Pain (Musculoskeletal and connective tissue disorders) | 13 (36) | 14 (29) — General Pain - not limited to a specific area
Elevation of liver function tests (Hepatobiliary disorders) | 3 (8) | 4 (12) — Elevated ALTs, ASTs or bilirubin was reported
Infection (Infections and infestations) | 13 (28) | 7 (17) — Infections included sinus infections, upper respiratory infections
Allergic (Endocrine disorders) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 15 (28) | 11 (16) — Most described as upset stomach, diarrhea, constipation
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 7 (12) — Described as shortness of breath
Edema/bruising (Blood and lymphatic system disorders) | 6 (9) | 7 (11) — Described as swelling in ankles and legs, increased bruising in the arms.
Ophthalomologic (Eye disorders) | 5 (5) | 4 (7) — Described as blurry vision
Dermatological (Skin and subcutaneous tissue disorders) | 3 (7) | 5 (10) — Described as dry skin
Constitutional/other (General disorders) | 10 (24) | 8 (34) — General fatigue
Muscle weakness/fatigue (Musculoskeletal and connective tissue disorders) | 10 (24) | 8 (34) — Worsening of the myasthenia gravis symptoms
Hematologic (Blood and lymphatic system disorders) | 6 (13) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No